CLINICAL TRIAL: NCT00092443
Title: Study of the Efficacy, Safety, and Immunogenicity of V260 at Expiry
Brief Title: Dose Confirmation Efficacy Study (V260-007)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V260-007; 2004_077
Record Dates: First submitted 2004-09-22; First posted 2004-09-27 (Estimated); Results first posted 2009-07-10 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-09

CONDITIONS: Rotavirus Infections
MeSH Terms: conditions — Rotavirus Infections | interventions — RotaTeq; Rotavirus Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- RotaTeq™ at Expiry Potency (≈1.1 x 10^7 IU/Dose) (Experimental): Three doses of RotaTeq™ (Rotavirus vaccine, live, oral, pentavalent)
  administered 28 to 70 days apart.
  Interventions: Biological: RotaTeq™, rotavirus vaccine, live, oral, pentavalent
- Placebo matching RotaTeq™ (Placebo Comparator): Placebo matching RotaTeq™ administered 28 to 70 days apart.
  Interventions: Biological: Comparator: Placebo matching RotaTeq™

INTERVENTIONS:
Biological: RotaTeq™, rotavirus vaccine, live, oral, pentavalent — Three doses of RotaTeq™ administered 28 to 70 days apart.
  Other Names: V260
  Arms: RotaTeq™ at Expiry Potency (≈1.1 x 10^7 IU/Dose)
Biological: Comparator: Placebo matching RotaTeq™ — Placebo matching RotaTeq™ administered 28 to 70 days apart.
  Arms: Placebo matching RotaTeq™

SUMMARY:
This study was designed to evaluate the safety of the investigational Rotavirus Vaccine and the efficacy to prevent Rotavirus Gastroenteritis.

DETAILED DESCRIPTION:
The duration of treatment is 10 months.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants

Exclusion Criteria:

* History of abdominal disorders from a birth defect, intussusception, or abdominal surgery
* Known or suspected problems with immune system
* Fever at time of immunization
* Prior administration of a rotavirus vaccine
* History of known prior rotavirus disease
* Chronic diarrhea, or failure to thrive

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1312 (Actual)
Dates: Start 2002-09; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Block SL, Vesikari T, Goveia MG, Rivers SB, Adeyi BA, Dallas MJ, Bauder J, Boslego JW, Heaton PM; Pentavalent Rotavirus Vaccine Dose Confirmation Efficacy Study Group. Efficacy, immunogenicity, and safety of a pentavalent human-bovine (WC3) reassortant rotavirus vaccine at the end of shelf life. Pediatrics. 2007 Jan;119(1):11-8. doi: 10.1542/peds.2006-2058. PMID 17200266

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 30 sites - 27 in the United States, and 3 in Finland from 24-Sep-2002 (first
  patient in) to 11-Feb-2004 (last dose given).
  Last subject completed follow-up: 08-Jun-2004.
  All data corrections applied (Frozen File): 07-Sep-2004
Pre-assignment Details: Excluded from the trial before assignment to groups were patients with: history of congenital abdominal
  disorders, intussusception, or abdominal surgery; history of known prior rotavirus disease, chronic diarrhea,
  or failure to thrive.
Groups:
- RotaTeq™ at Expiry Potency (≈1.1 x 10^7 IU/Dose): Three doses of RotaTeq™ (Rotavirus vaccine, live, oral, pentavalent) administered 28 to 70 days apart, with up to 42 days of safety follow-up after each vaccination, and followup for acute gastrointestinal episodes (AGEs) through the first rotavirus season post vaccination.
- Placebo Matching RotaTeq™: Placebo matching RotaTeq™ administered 28 to 70 days apart, with up to 42 days of safety follow-up after each vaccination and follow-up for acute gastrointestinal episodes (AGEs) through the first rotavirus season post vaccination.
Period: Overall Study
Arm/Group | RotaTeq™ at Expiry Potency (≈1.1 x 10^7 IU/Dose) | Placebo Matching RotaTeq™
Started | 651 (Subjects who passed all entry criteria and who were randomized in to the study) | 661 (Subjects who passed all entry criteria and who were randomized in to the study)
Vaccinated at Visit 1 | 650 | 660
Vaccinated at Visit 2 | 618 | 627
Vaccinated at Visit 3 | 593 | 608
Completed | 593 (Subjects vaccinated and followed up 42 days after each dose, thru 1st rotavirus season post study) | 607 (Subjects vaccinated and followed up 42 days after each dose, thru 1st rotavirus season post study)
Not Completed | 58 | 54
Not completed — Adverse Event | 9 | 13
Not completed — Lost to Follow-up | 7 | 3
Not completed — Protocol Violation | 11 | 9
Not completed — Withdrawal by Subject | 9 | 11
Not completed — Moved | 5 | 5
Not completed — Other | 17 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RotaTeq™ at Expiry Potency (≈1.1 x 10^7 IU/Dose) | Placebo Matching RotaTeq™ | Total
Number analyzed (Participants) | 651 | 661 | 1312
Age, Customized [Number; unit: participants]
  6 to 12 Weeks | 648 | 658 | 1306
  Over 12 Weeks | 3 | 3 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 304 | 323 | 627
  Male | 347 | 338 | 685
Race/Ethnicity [Number; unit: participants]
  White | 525 | 540 | 1065
  Hispanic American | 79 | 77 | 156
  Black | 21 | 23 | 44
  Multi-Racial | 17 | 15 | 32
  Other | 9 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Occurence of Clinical Rotavirus Disease Caused by the Composite of the Serotypes Contained Within the Vaccine More Than 14 Days Following the Third Dose.
Description: G1, G2, G3, and G4 Serotype Rotavirus Gastroenteritis Cases Occurring at Least 14 Days Postdose 3 Through the First Rotavirus Season Postvaccination in the Per-Protocol Population Using Per-Protocol Case Definition
Time Frame: At least 14 days following the 3rd vaccination
Population: Per Protocol Population; number randomized is different from number analyzed due to some data excluded from the analysis (e.g., unevaluable due to wild-type rotavirus-positive stool antigen Enzyme immunoassay (EIA) prior to 14 days Postdose 3, incomplete clinical and/or laboratory results, or stool samples collected out of day range.
Measure: Number; unit: Participants
Groups:
- RotaTeq™ at Expiry Potency (≈1.1 x 107 IU/Dose): Three doses of RotaTeq™ (Rotavirus vaccine, live, oral, pentavalent) administered 28 to 70 days apart, with up to 42 days of safety follow-up after each vaccination, and follow-up for acute gastrointestinal episodes (AGEs) through the first rotavirus season post vaccination.
- Placebo Matching RotaTeq™: Placebo matching RotaTeq™ administered 28 to 70 days apart, with up to 42 days of safety follow-up after each vaccination and follow-up for AGEs through the first rotavirus season post vaccination.
Arm/Group | RotaTeq™ at Expiry Potency (≈1.1 x 107 IU/Dose) | Placebo Matching RotaTeq™
Number analyzed (Participants) | 551 | 564
Participants | 15 | 54
Statistical Analysis 1: Comparison: RotaTeq™ at Expiry Potency (≈1.1 x 107 IU/Dose) vs Placebo Matching RotaTeq™; Test type: Superiority or Other; p < 0.001, Exact Binomial Test; Efficacy = 1-Relative Risk = 72.5, 95% CI [50.6 to 85.6] — Efficacy = 1-RR, expressed as a percentage; the RR is the incidence in the vaccine group / the incidence in the placebo group

2. Secondary Outcome: Number of Subjects With ≥3 Fold Rise in Antibody Titer
Description: Induction of postdose 3 rotavirus Serum neutralizing antibody (SNA) response (Number of subjects with ≥3 fold rise in antibody titer)
Time Frame: 14 days following the 3rd vaccination
Population: Per Protocol Population; number randomized is different from number analyzed due to some data excluded from the analysis (e.g., unevaluable due to wild-type rotavirus-positive stool antigen EIA prior to 14 days Postdose 3, incomplete clinical and/or laboratory results, or stool samples collected out of day range.
Measure: Number; unit: Participants
Groups:
- RotaTeq™ at Expiry Potency (SNA - G1); RotaTeq™ at Expiry Potency (SNA - G2); RotaTeq™ at Expiry Potency (SNA - G3); RotaTeq™ at Expiry Potency (SNA - G4); RotaTeq™ at Expiry Potency (SNA - P1A); Placebo Matching RotaTeq™ (SNA - G1); Placebo Matching RotaTeq™ (SNA - G2); Placebo Matching RotaTeq™ (SNA - G3); Placebo Matching RotaTeq™ (SNA - G4); Placebo Matching RotaTeq™ (SNA - P1A): Subjects tested with data available for analysis excluding protocol violators and subjects with invalid data based on lab determinations.
Arm/Group | RotaTeq™ at Expiry Potency (SNA - G1) | RotaTeq™ at Expiry Potency (SNA - G2) | RotaTeq™ at Expiry Potency (SNA - G3) | RotaTeq™ at Expiry Potency (SNA - G4) | RotaTeq™ at Expiry Potency (SNA - P1A) | Placebo Matching RotaTeq™ (SNA - G1) | Placebo Matching RotaTeq™ (SNA - G2) | Placebo Matching RotaTeq™ (SNA - G3) | Placebo Matching RotaTeq™ (SNA - G4) | Placebo Matching RotaTeq™ (SNA - P1A)
Number analyzed (Participants) | 67 | 62 | 67 | 63 | 61 | 73 | 70 | 75 | 70 | 69
Participants | 38 | 9 | 6 | 25 | 15 | 2 | 0 | 0 | 1 | 2
Statistical Analysis 1: Comparison: RotaTeq™ at Expiry Potency (SNA - G1); Test type: Superiority or Other; Percent of Participants = 56.7, 95% CI [44.0 to 66.8]
Statistical Analysis 2: Comparison: Placebo Matching RotaTeq™ (SNA - G1); Test type: Superiority or Other; Percent of Participants = 2.7, 95% CI [0.3 to 9.5]
Statistical Analysis 3: Comparison: RotaTeq™ at Expiry Potency (SNA - G2); Test type: Superiority or Other; Percent of Participants = 14.5, 95% CI [6.9 to 25.8]
Statistical Analysis 4: Comparison: Placebo Matching RotaTeq™ (SNA - G2); Test type: Superiority or Other; Percent of Participants = 0.0, 95% CI [0.0 to 5.1]
Statistical Analysis 5: Comparison: RotaTeq™ at Expiry Potency (SNA - G3); Test type: Superiority or Other; Percent of Participants = 9.0, 95% CI [3.4 to 18.5]
Statistical Analysis 6: Comparison: Placebo Matching RotaTeq™ (SNA - G3); Test type: Superiority or Other; Percent of Participants = 0.0, 95% CI [0.0 to 4.8]
Statistical Analysis 7: Comparison: RotaTeq™ at Expiry Potency (SNA - G4); Test type: Superiority or Other; Percent of Participants = 39.7, 95% CI [27.6 to 52.8]
Statistical Analysis 8: Comparison: Placebo Matching RotaTeq™ (SNA - G4); Test type: Superiority or Other; Percent of Participants = 1.4, 95% CI [0.0 to 7.7]
Statistical Analysis 9: Comparison: RotaTeq™ at Expiry Potency (SNA - P1A); Test type: Superiority or Other; Percent of Participants = 24.6, 95% CI [14.5 to 37.3]
Statistical Analysis 10: Comparison: Placebo Matching RotaTeq™ (SNA - P1A); Test type: Superiority or Other; Percent of Participants = 2.9, 95% CI [0.4 to 10.1]

ADVERSE EVENTS:
Groups:
- RotaTeq™ at Expiry Potency (≈1.1 x 10^7 IU/Dose): Three doses of RotaTeq™ (Rotavirus vaccine, live, oral, pentavalent) administered 28 to 70 days apart, with up to 42 days of safety follow-up after each vaccination, and follow-up for acute gastrointestinal episodes (AGEs) through the first rotavirus season post vaccination.
Arm/Group | RotaTeq™ at Expiry Potency (≈1.1 x 10^7 IU/Dose) | Placebo Matching RotaTeq™
Serious Adverse Events (participants affected / at risk) | 21/649 | 28/658
Other Adverse Events (participants affected / at risk) | 558/649 | 565/658
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RotaTeq™ at Expiry Potency (≈1.1 x 10^7 IU/Dose) (N=649) | Placebo Matching RotaTeq™ (N=658)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Perirectal abscess (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Sudden infant death syndrome (General disorders) | 1 (1) | 0 (0)
Milk allergy (Immune system disorders) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 7 (7) | 7 (7)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Croup infectious (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 2 (2)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Pertussis (Infections and infestations) | 0 (0) | 3 (3)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 2 (2)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 1 (1)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral cyst (Nervous system disorders) | 0 (0) | 1 (1)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RotaTeq™ at Expiry Potency (≈1.1 x 10^7 IU/Dose) (N=649) | Placebo Matching RotaTeq™ (N=658)
Conjunctivitis (Eye disorders) | 50 (56) | 46 (53)
Constipation (Gastrointestinal disorders) | 35 (39) | 34 (38)
Diarrhoea (Gastrointestinal disorders) | 103 (160) | 110 (177)
Flatulence (Gastrointestinal disorders) | 52 (72) | 49 (78)
Regurgitation of food (Gastrointestinal disorders) | 44 (54) | 41 (55)
Vomiting (Gastrointestinal disorders) | 81 (112) | 77 (116)
Injection site pain (General disorders) | 61 (82) | 62 (81)
Pyrexia (General disorders) | 283 (450) | 265 (438)
Gastroenteritis (Infections and infestations) | 91 (103) | 106 (132)
Otitis media (Infections and infestations) | 119 (143) | 111 (144)
Respiratory tract infection (Infections and infestations) | 41 (46) | 28 (32)
Rhinitis (Infections and infestations) | 69 (84) | 81 (110)
Upper respiratory tract infection (Infections and infestations) | 150 (192) | 143 (172)
Agitation (Psychiatric disorders) | 102 (145) | 99 (145)
Crying (Psychiatric disorders) | 53 (82) | 52 (79)
Irritability (Psychiatric disorders) | 155 (248) | 172 (299)
Cough (Respiratory, thoracic and mediastinal disorders) | 95 (111) | 90 (106)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 39 (47) | 53 (68)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 59 (73) | 42 (50)

LIMITATIONS AND CAVEATS:
Safety has been reported in the literature.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.